CLINICAL TRIAL: NCT02832141
Title: Effect of Thoracic Spine Mobilization on Skin-blood Flow, Erythema and Sympathetic Nervous Systems
Brief Title: Effect of Thoracic Spine Mobilization on Sympathetic Nervous Systems
Status: Completed | Type: Observational
Sponsor: Bern University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Slavko Rogan, MSc, MA, Bern University of Applied Sciences
Other Study IDs: Mobilization Thoracic Spine
Record Dates: First submitted 2016-07-02; First posted 2016-07-14 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Erythema
Keywords: Skin blood flow; Skin redness; Sympathetic nervous system; Regional Blood Flow
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Group A: immediate effects: T0, Grade 3 central thoracic mobilization from posterior-to-anterior on thoracic vertebrae from T5 to T12, immediate (T1), after 2 (T2), 4 (T3), 6 (T4), 8 (T5) and 10 (T6) minutes, 1 days wash-out period; T7, a grade 3 central thoracic mobilization from anterior-to-posterior on all thoracic vertebrae, immediate T8, after 2 (T9), 4 (T10), 6 (T11), 8 (T12) and 10 (T13) minutes.
  Interventions: Procedure: Mobilization anterior; Procedure: Mobilization posterior
- Group B: Group B: immediate effects: T0, 3 central thoracic mobilization from anterior-to-posterior on thoracic vertebrae from T5 to T12, immediate (T1), after 2 (T2), 4 (T3), 6 (T4), 8 (T5) and 10 (T6) minutes, 1 days wash-out period; T7, a grade 3-4 central thoracic mobilization from posterior-to-anterior on all thoracic vertebrae, immediate T8, after 2 (T9), 4 (T10), 6 (T11), 8 (T12) and 10 (T13) minutes.
  Interventions: Procedure: Mobilization anterior; Procedure: Mobilization posterior

INTERVENTIONS:
Procedure: Mobilization anterior — Participant in prone position. Central thoracic mobilization from posterior-to-anterior.
  Other Names: Thoracic spine mobilization with anterior pressure
Procedure: Mobilization posterior — Participant in sitting position. Central thoracic mobilization from anteriors-to-posterior.
  Other Names: Thoracic spine mobilization with posterior pressure

SUMMARY:
This pilot study aims to i) represents the feasibility of the study design and ii) to point out acute effects of thoracic spine mobilization on skin-blood flow, erythema and the sympathetic nervous system.

ELIGIBILITY:
Inclusion Criteria:

* age 20 - 30 years
* healthy persons

Exclusion Criteria:

* current pain
* blood pressure medications
* osteoporosis
* cardiac or neurological symptoms
* pregnancy
* thromobosis

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy person between 20 and 30 years.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility: Adherence of recruited participants | Every 4 weeks up to 2 years
  Defined as the number of drop-outs and presence of participants which invited. Measurement unit: number
Feasibility of the investigating procedure | Every 4 weeks up to 2 years
  Measured the burden of testing procedure. Measurement units = number and percentage
Feasibility of the mobilization intervention from posterior-to-anterior on thoracic vertebrae | Every 4 weeks up to 2 years
  Measured adverse effects as pain and harm results to participants. Measurement units = number and percentage
Feasibility of the mobilization intervention from anterior-to-posterior on thoracic vertebrae | Every 4 weeks up to 2 years
  Measured as adverse effects as pain and harm results to participants. Measurement units = number and percentage.

SECONDARY OUTCOMES:
Rate of heart rate variability (HRV) | Change from baseline imediately after, 2, 4, 6, 8 and 10 minutes after the intervention
  HRV is measured as the variations of the time interval between two consecutive cardiac beats registered by means Polar watch RS800 is used to measures (HRV). Measurement unit: High frequency-band (HF-Band) and Low frequency-band (LF-Band)
Rate of systolic blood pressure value (mmHg) | Change from baseline imediately after, 2, 4, 6, 8 and 10 minutes after the intervention
  Omron MIT Elite Plus is used for measuring systolic blood flow. iMeasurement units: mmHg (millimeter of mercury)
Rate of diastolic blood pressure value (mmHg) changes | Change from baseline imediately after, 2, 4, 6, 8 and 10 minutes after the intervention
  Omron MIT Elite Plus is used for measuring diastolic blood pressureMeasurement units: mmHg (millimeter of mercury)
Rate of heartbeat frequency | Change from baseline imediately after, 2, 4, 6, 8 and 10 minutes after the intervention
  Polar watch RS800 is used for measuring heartbeat frequency. Measurement units: beat per minute (bpm)
Rate of skin-blood flow variation | Change from baseline imediately after, 2, 4, 6, 8 and 10 minutes after the intervention
  Laser doppler imaging is used for measuring microcirculatory changes. Measurement units: perfusion unit
Rate of erythema | Change from baseline imediately after, 2, 4, 6, 8 and 10 minutes after the intervention
  Tristimulus surface colorimetry is used for measuring erythema. Measurement units: Erythema index

CONTACTS AND LOCATIONS:
Overall Officials: Jan Taeymans, PhD, Principal Investigator — Bern University of Applied Science, Departement Health
Locations (1):
- Bern University of Applied Science, Department Health, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rogan S, Taeymans J, Clarys P, Clijsen R, Tal-Akabi A. Feasibility and effectiveness of thoracic spine mobilization on sympathetic/parasympathetic balance in a healthy population - a randomized controlled double-blinded pilot study. Arch Physiother. 2019 Dec 9;9:15. doi: 10.1186/s40945-019-0067-2. eCollection 2019. PMID 31867125